CLINICAL TRIAL: NCT06778486
Title: CHAT-OA: Conversations in Health Literacy Using AI Technology for Osteoarthritis Patients
Brief Title: Conversations in Health Literacy Using AI Technology for Osteoarthritis Patients
Acronym: CHAT-OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2169004
Record Dates: First submitted 2024-11-22; First posted 2025-01-16 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis; Osteoarthritis of the Hip or Knee
Keywords: artificial intelligence; health literacy; decisional conflict
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): This arm will undergo standard clinical care without the intervention.
- Artificial Intelligence Chatbot (Experimental): This arm will interact with an artificial intelligence chatbot prior to their clinic visit.
  Interventions: Other: Artificial Intelligence Chatbot

INTERVENTIONS:
Other: Artificial Intelligence Chatbot — The intervention is a generative artificial intelligence large language model chatbot that has a structured prompt with fill-in-the-blank style questions that the participant will complete.
  Arms: Artificial Intelligence Chatbot

SUMMARY:
The goal of this clinical trial is to assess the use of a generative artificial intelligence large language model chatbot in improving decision making factors in patients with hip and knee osteoarthritis. The main questions it aims to answer are:

Does the use of an artificial intelligence chatbot have an effect on decisional conflict and anxiety related to decision making? Are changes in decisional conflict correlated with changes in patient reported outcomes? Are changes in decisional conflict correlated with health literacy? Participants will interact with an artificial intelligence chatbot prior to their clinic visit with an orthopaedic surgeon, using a structured prompt.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Ability to read and write in English
* All races and ethnicities
* Clinical symptoms of hip and/or knee osteoarthritis

Exclusion Criteria:

* Inability to read and write in English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale | At three time points: Within one week after the clinic visit, 1 month after the clinic visit, 6 months after the clinic visit.
  16 questions with Likert scale style answers ranging from 0 to 4. The raw score is converted to a score out of 100. The score ranges from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
Beck Anxiety Inventory | At three time points: Within one week after the clinic visit, 1 month after the clinic visit, 6 months after the clinic visit.
  21 questions with Likert scale style answers ranging from 0 to 4. The raw score is the sum of the answers, which is converted to a score out of 100. The score ranges from 0 (low anxiety) to 63 (high anxiety).

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score for Joint Replacement | At enrollment
  7 questions with Likert scale style answers ranging from 0 to 4. The raw score is the sum of the answers, which is converted to a score out of 100. The score ranges from 0 (total knee disability) to 100 (perfect knee health).
Hip dysfunction and Osteoarthritis Outcome Score for Joint Replacement | At enrollment
  6 questions with Likert scale style answers ranging from 0 to 4. The raw score is the sum of the answers, which is converted to a score out of 100. The score ranges from 0 (total hip disability) to 100 (perfect hip health).
Patient-Reported Outcomes Measurement Information System Global Health Version 1.2 | At enrollment
  10 questions with Likert scale style answers ranging from 1 to 5 and 1 question about pain with answers from 0 to 10. The questions are grouped into 4 sub-groups corresponding to physical and mental health main groups, in addition to the pain score. The raw scores are a sum of the answers for both physical and mental health range from 4 (poor physical or mental health) to 20 (best possible physical or mental health). The raw score is then converted to a t-score using the associated tables with the range 16.2 (worst possible physical or mental health) to 67.7 (best possible physical or mental health). The t-score is interpreted in comparison to the general population that has a mean of 50 and standard deviation of 10.

OTHER OUTCOMES:
Visual Analog Scale Pain Score | At enrollment
  3 questions evaluating pain and different time points, each with answers ranging from 0 (no pain) to 100 (worst pain imaginable).
Health Literacy Single Item Screener | At enrollment
  Both questions 1 and 2 have Likert scale style answers from 1 (limited ability to navigate healthcare scenarios independently) to 5 (adequate ability to navigate healthcare scenarios independently).
Newest Vital Sign | At enrollment
  This measure involves participants answering a series of questions based on their interpretation of a nutrition label. It includes 5 primary questions with an additional conditional question, making up to 6 questions in total, depending on the participant's responses. This assessment is designed to evaluate health literacy, specifically the ability to understand and apply nutritional information. The score is the sum of the correct answers, ranging from 0 (indicating limited health literacy) to 6 (indicating adequate health literacy).
Literacy in Musculoskeletal Problems | At enrollment
  9 questions each with 4 answers, in addition to an "I don't know" selection. The total score is the sum of the correct answers ranging from 0 (poor musculoskeletal health literacy) to 9 (excellent musculoskeletal health literacy).
Rapid Estimate of Adult Literacy in Medicine - Short Form | At the first clinic visit after enrollment
  7-item word recognition test to provide clinicians with a valid quick assessment of patient health literacy. The test is administered in-person by a clinician. The participant is given a list of words by a clinician and asked to pronounce the words. The clinician listens and evaluates the number of words the participant pronounces correctly and the total score is based on the number of words that are correctly pronounced. A higher score is indicative of higher health literacy. The maximum score of 7 is correlated with high health literacy equivalent to high school education or greater, and a participants ability to read most patient education materials. The minimum score of 0 is associated with low health literacy equivalent to third grade education or below, and a participants inability to read most low-literacy patient education materials.
Flesch-Kincaid Readability Test | Within 1 month of AI chatbot use
  This test will be used to evaluate the readability of the chatbot outputs that are presented to the participants, and will be conducted by an investigator. This test analyzes free text and determines a readability score ranging from 0 (very difficult to read) to 100 (very easy to read), and corresponds to the education level required to read the text.
Simple Measure of Gobbleygook | Within 1 month of AI chatbot use
  This test will be used to evaluate the readability of the chatbot outputs that are presented to the participants and it will be conducted by an investigator. This test analyzes free text and determines a readability score with a minimum of 4.1721 and a maximum that is theoretically infinite. The number of the score is equivalent to the approximate school grade level required to read the text.
5-point Likert Safety-Harm Scale | Within 1 week of AI chatbot use
  This safety evaluation tool will be used by a physician to assess chatbot outputs that are presented to the participant with a Likert scale ranging from 0 (no likelihood of harm) to 5 (high likelihood of harm).

CONTACTS AND LOCATIONS:
Overall Officials: Zachary C Lum, DO, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No